CLINICAL TRIAL: NCT07285213
Title: A Phase IIb, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of AZD5148 for Prevention of Recurrence of Clostridioides Difficile Infection in Individuals 18 Years of Age and Above
Brief Title: Prevention of Recurrent C. Difficile Infection Study With AZD5148 Monoclonal Antibody
Acronym: PRISM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D8820C00003
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides Difficile infection; C. Diff; CDiff; Clostridiodes Difficile Infection prevention of recurrence
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD5148: dose A (Experimental): Participants will receive a single dose A of AZD5148 administered via either intramuscular injection or intravenous push.
  Interventions: Drug: AZD5148
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo via intramuscular or intravenous push.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD5148 — Participants will receive a single dose A of AZD5148 administered via either intramuscular injection or intravenous push.
  Arms: AZD5148: dose A
Other: Placebo — Participants will receive a single dose of placebo (0.9% (w/v) sodium chloride for injection) administered via either intramuscular injection or intravenous push.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AZD5148 for prevention of recurrence of Clostridioides difficile infection in Individuals 18 years of age and above.

DETAILED DESCRIPTION:
Approximately 230 participants will be enrolled and randomized 1:1 to receive a single dose of either AZD5148 or placebo (normal saline). Route of administration (intramuscular or intravenous push) will be according to the Investigator's choice. Stratification will be based on geographical region.

Study details include:

* Up to 2 site visits for confirmation of eligibility and dose administration, including stool sample collection;
* Up to 7 planned visits;
* Contacts initiated by site staff -weekly, later monthly follow up;
* Electronic diary completion.

ELIGIBILITY:
Inclusion Criteria:

Participant must be ≥ 18 years of age at the time of signing the informed consent, capable of giving signed informed consent.

Participants with a qualifying C. difficile infection episode at the time of providing informed consent defined by:

* Positive local C. difficile toxin test (eg, immune assay or CCNA) on an unformed stool sample collected during this episode, and
* Receipt of standard of care antibacterial drug therapy for C. difficile infection (fidaxomicin, vancomycin or metronidazole) for this episode, with planned duration of at least 10 and at most 25 days at time of IMP administration.

Note: Diarrhea is not required to be present on the day of investigational medicinal product (IMP) administration.

Body weight ≥ 40 kg

Exclusion Criteria:

History of inflammatory bowel disease (eg, ulcerative colitis, Crohn's disease, microscopic colitis).

Participant with a non - CDI (C. difficile infection) condition such that the participant routinely passes loose stool (eg, patients with an ostomy)

Planned surgery for C. difficile infection within 24 hours of enrollment

Current toxic megacolon and/or small bowel ileus

Any history of total colectomy or bariatric surgery (bariatric surgery which does not disrupt the gastrointestinal lumen, ie, restrictive procedures such as banding, are permitted).

Major gastrointestinal surgery as assessed by the Investigator (eg, significant bowel resection or diversion) within 90 days before enrollment (this does not include appendectomy or cholecystectomy)

Due to receive more than 25 days of antibacterial drug therapy for C. difficile infection for the qualifying C. difficile infection episode

Treatment with a fecal donor transplant or fecal microbiota product in the 180 days before IMP administration, are receiving or planned administration for the qualifying episode of C. difficile infection, or planned administration during the 180 days after IMP administration

Treatment with bezlotoxumab in the 180 days before IMP administration, are receiving or planned administration for the qualifying episode of CDI, or planned administration during the 180 days after IMP administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-04-20 (Estimated); Study Completion 2028-01-18 (Estimated)

PRIMARY OUTCOMES:
First occurrence of recurrence of C difficile infection | Day 1 through day 91
  rCDI is a recurrence of C difficile infection (CDI) occurring after initial clinical cure of the qualifying CDI. CDI is defined as a history of diarrhea (>=3 unformed stools, ie, type 6 or 7 stool on Bristol Stool Scale in <=24 hours for 2 consecutive calendar days) accompanied by a positive stool test for C difficile toxin.

SECONDARY OUTCOMES:
Sustained clinical cure | Day 91
  Sustained clinical cure is defined as achieving initial clinical cure (ICC) of the qualifying CDI and not having an rCDI event through Day 91. ICC is defined as clinical cure for the qualifying CDI episode with a duration of a minimum of 10 days and a maximum of 25 days of standard of care antibacterial drug therapy for CDI.
Duration of recurrent C difficile infection | Day 1 through Day 91
  Duration of the first occurrence of confirmed rCDI is calculated from the first day of diarrhea meeting the clinical symptom criteria until the date of clinical cure. Clinical cure is defined as <=2 unformed stools (ie, type 6 or 7 stool on Bristol Stool Scale) in 24 hours for 2 consecutive calendar days after the end of antibacterial drug treatment for the CDI episode.
First occurrence of severe recurrent C difficile infection | Day 1 through Day 91
  Severe rCDI is defined as an rCDI event characterized by either: peripheral blood leukocytosis with leukocyte count >15,000 cells/uL or serum creatinine level >1.5 mg/dL.
First occurrence of fulminant recurrent C difficile infection | Day 1 through Day 91
  Fulminant rCDI is defined as a severe rCDI event with hypotension or shock, toxic megacolon, or ileus.
Severity of participant reported diarrhea symptoms | Day 1 through Day 91
  As reported by patient reported outcome (PRO) instrument for first occurrence of rCDI.
Duration of participant reported diarrhea symptoms | Day 1 through Day 91
  As reported by patient reported outcome (PRO) instrument for first occurrence of rCDI.
Occurrence of recurrent C difficile related mortality | Day 1 through Day 91
  rCDI related mortality is defined as a death related to rCDI as assessed by the Investigator.
Immediate adverse events | 1 hour post-IMP administration
  Adverse events with a start time within 1 hour post-IMP administration
Injection/Infusion-related reactions | 24 hours post-IMP administration
  Injection or infusion-related reactions with a start date and time within 24 hours of IMP administration.
Local reactions at the injection/infusion site | Day 1 through Day 8
  Local reactions at the injection or infusion site with a start date through Day 8 post-IMP administration.
Serious adverse events | ICF date through Day 361
  SAEs are adverse events that fulfill any of the SAE criteria and are recorded with a start date from the date of informed consent form signature until the end of the study follow-up (Day 361)
Medically attended adverse events (MAAEs) | Day 1 through Day 361
  MAAEs are adverse events leading to medically attended visits that were not routine visits, such as ER visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason.
Adverse events of special interest (AESIs) | Day 1 through Day 361
  AESIs as defined by Clinical Study Protocol.
Related adverse events | Day 1 through Day 361
  Related AEs are adverse events assessed as related to IMP by the Investigator.
Adverse events | Day 1 through Day 91
  AEs are defined as any unfavourable medical occurrence in a participant administered the IMP, regardless of the causal relationship to IMP.
Pharmacokinetics of AZD5148 | Day 1 through Day 361
  PK will be characterized through AZD5148 serum concentrations over time in participants who receive AZD5148.
Anti-drug antibodies to AZD5148 | Day 1 through Day 361
  Immunogenicity is evaluated through AZD5148 anti-drug antibody responses over time in serum from participants who receive AZD5148.

CONTACTS AND LOCATIONS:
Locations (104):
- United States (38):
  - Research Site, Phoenix, Arizona
  - Research Site, Chula Vista, California
  - Research Site, Sacramento, California
  - Research Site, Torrance, California
  - Research Site, Hamden, Connecticut
  - Research Site, Gainesville, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Miramar, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Burr Ridge, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Potomac, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Hartsdale, New York
  - Research Site, Inwood, New York
  - Research Site, The Bronx, New York
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Johnson City, Tennessee
  - Research Site, Charlottesville, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Australia (5):
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, Herston
  - Research Site, Melbourne
  - Research Site, South Brisbane
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hvidovre
  - Research Site, København Ø
  - Research Site, Odense C
- France (6):
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Tours
- Germany (8):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Leipzig
  - Research Site, München
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Thessaloniki
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Kistarcsa
  - Research Site, Pécs
- Italy (6):
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Varese
- Japan (6):
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Meguro-ku
  - Research Site, Nagasaki
  - Research Site, Shimonoseki-shi
  - Research Site, Yaizu-shi
- Poland (2):
  - Research Site, Lublin
  - Research Site, Warsaw
- Spain (5):
  - Research Site, Alicante
  - Research Site, Badalona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
- Sweden (4):
  - Research Site, Helsingborg
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Västerås
- United Kingdom (2):
  - Research Site, Birmingham
  - Research Site, Cambridge

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/